CLINICAL TRIAL: NCT03326297
Title: Effectiveness of Manual Therapy Through Osteopathy in the Treatment of Infant Colic.
Brief Title: Physiotherapy and Osteopathy on Infant Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-0021-2015
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Infantile Colic; Manual Therapy
Keywords: Infant Colic; Osteopathy; Stress; Physiotherapy
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteopathy manual therapy (Experimental): Osteopathy manual therapy applying the following treatment: Technique for the treatment of parasympathetic innervation, Techniques for the treatment of sympathetic innervation of the digestive system, Functional visceral techniques.
  Interventions: Other: Osteopathy manual therapy
- Measures to support and education to the family (Active Comparator): Measures to support and education to the family that consist on pedagogical intervention in parents, health education.
  Interventions: Behavioral: Measures to support and education to the family
- No specific intervention (No Intervention): No specific intervention, prescriptions by pediatrician

INTERVENTIONS:
Other: Osteopathy manual therapy — Technique for the treatment of parasympathetic innervation, Techniques for the treatment of sympathetic innervation of the digestive system, Functional visceral techniques.
  Arms: Osteopathy manual therapy
Behavioral: Measures to support and education to the family — Pedagogical intervention in parents and health education
  Arms: Measures to support and education to the family

SUMMARY:
This study compares the effectiveness of manual therapy (osteopathy) on infant colic versus education to the family, and a third group with no specific intervention.

DETAILED DESCRIPTION:
Infant colic is a problem that affects 10-30% of babies in their first months of life. This research project aims to verify the effectiveness of manual therapy on infant colic. The sample is divided in three groups, performing in the firts one osteopathy manual therapy; in the second one, measures to support and education to the family; and in the third, there is no specific intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed if Infant Colic.

Exclusion Criteria:

* Babies diagnosed of other pathologies that justify cries, such as reflux, food intolerances or neurological syndromes.
* Premature babies less than 37 weeks gestation, who may be involved in other concomitant pathologies.
* Mothers (families) with language barriers, due to the difficulty of collecting data.

Ages: 3 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline FCL Questionnaire at 12 weeks of infants' life. | At baseline, at 4 weeks, at 8 weeks, at 12 weeks of infants' life and at 3 months of infants' life
  FCL (Fisioterapia en el Cólico del Lactante) QUESTIONNAIRE: Infant colic assessment questionnaire. Group CTS (Ciencias y Técnicas de la Salud) 305 of the University of Seville.

SECONDARY OUTCOMES:
Maternal stress in the last month. | At baseline and at 12 weeks of infants' life.
  Perceived Stress Questionnaire (PSQ).
Intensity of irritability | At baseline and at 12 weeks of infants' life
  Analogue visual scale from 0 to 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain

REFERENCES:
- [Background] Gudmundsson G. Infantile colic: is a pain syndrome. Med Hypotheses. 2010 Dec;75(6):528-9. doi: 10.1016/j.mehy.2010.07.014. Epub 2010 Aug 21. PMID 20729004
- [Background] Kim JS. Acute abdominal pain in children. Pediatr Gastroenterol Hepatol Nutr. 2013 Dec;16(4):219-24. doi: 10.5223/pghn.2013.16.4.219. Epub 2013 Dec 31. PMID 24511517
- [Background] Cohen-Silver J, Ratnapalan S. Management of infantile colic: a review. Clin Pediatr (Phila). 2009 Jan;48(1):14-7. doi: 10.1177/0009922808323116. Epub 2008 Oct 2. PMID 18832537
- [Background] Akman I, Kuscu K, Ozdemir N, Yurdakul Z, Solakoglu M, Orhan L, Karabekiroglu A, Ozek E. Mothers' postpartum psychological adjustment and infantile colic. Arch Dis Child. 2006 May;91(5):417-9. doi: 10.1136/adc.2005.083790. Epub 2006 Feb 1. PMID 16452109
- [Background] Alcantara J, Alcantara JD, Alcantara J. The chiropractic care of infants with colic: a systematic review of the literature. Explore (NY). 2011 May-Jun;7(3):168-74. doi: 10.1016/j.explore.2011.02.002. PMID 21571236
- [Background] Miller-Loncar C, Bigsby R, High P, Wallach M, Lester B. Infant colic and feeding difficulties. Arch Dis Child. 2004 Oct;89(10):908-12. doi: 10.1136/adc.2003.033233. PMID 15383432
- [Background] Anabrees J, Indrio F, Paes B, AlFaleh K. Probiotics for infantile colic: a systematic review. BMC Pediatr. 2013 Nov 15;13:186. doi: 10.1186/1471-2431-13-186. PMID 24238101
- [Background] Levitzky S, Cooper R. Infant colic syndrome--maternal fantasies of aggression and infanticide. Clin Pediatr (Phila). 2000 Jul;39(7):395-400. doi: 10.1177/000992280003900703. PMID 10914303
- [Background] Hall B, Chesters J, Robinson A. Infantile colic: a systematic review of medical and conventional therapies. J Paediatr Child Health. 2012 Feb;48(2):128-37. doi: 10.1111/j.1440-1754.2011.02061.x. Epub 2011 Apr 7. PMID 21470331
- [Background] Sung V, Collett S, de Gooyer T, Hiscock H, Tang M, Wake M. Probiotics to prevent or treat excessive infant crying: systematic review and meta-analysis. JAMA Pediatr. 2013 Dec;167(12):1150-7. doi: 10.1001/jamapediatrics.2013.2572. PMID 24100440
- [Background] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Background] Tekgunduz KS, Gurol A, Apay SE, Caner I. Effect of abdomen massage for prevention of feeding intolerance in preterm infants. Ital J Pediatr. 2014 Nov 14;40:89. doi: 10.1186/s13052-014-0089-z. PMID 25394549
- [Background] Savino F, Ceratto S, De Marco A, Cordero di Montezemolo L. Looking for new treatments of Infantile Colic. Ital J Pediatr. 2014 Jun 5;40:53. doi: 10.1186/1824-7288-40-53. PMID 24898541
- [Background] Skjeie H, Skonnord T, Fetveit A, Brekke M. Acupuncture for infantile colic: a blinding-validated, randomized controlled multicentre trial in general practice. Scand J Prim Health Care. 2013 Dec;31(4):190-6. doi: 10.3109/02813432.2013.862915. Epub 2013 Nov 15. PMID 24228748
- [Background] Savino F, Tarasco V. New treatments for infant colic. Curr Opin Pediatr. 2010 Dec;22(6):791-7. doi: 10.1097/MOP.0b013e32833fac24. PMID 20859207
- [Background] Ernst E. Chiropractic treatment for gastrointestinal problems: a systematic review of clinical trials. Can J Gastroenterol. 2011 Jan;25(1):39-40. doi: 10.1155/2011/910469. PMID 21258667
- [Background] Wiberg KR, Wiberg JM. A retrospective study of chiropractic treatment of 276 danish infants with infantile colic. J Manipulative Physiol Ther. 2010 Sep;33(7):536-41. doi: 10.1016/j.jmpt.2010.08.004. PMID 20937431
- [Background] Miller JE, Newell D, Bolton JE. Efficacy of chiropractic manual therapy on infant colic: a pragmatic single-blind, randomized controlled trial. J Manipulative Physiol Ther. 2012 Oct;35(8):600-7. doi: 10.1016/j.jmpt.2012.09.010. PMID 23158465
- [Background] Miller JE, Phillips HL. Long-term effects of infant colic: a survey comparison of chiropractic treatment and nontreatment groups. J Manipulative Physiol Ther. 2009 Oct;32(8):635-8. doi: 10.1016/j.jmpt.2009.08.017. PMID 19836599
- [Background] Olafsdottir E, Forshei S, Fluge G, Markestad T. Randomised controlled trial of infantile colic treated with chiropractic spinal manipulation. Arch Dis Child. 2001 Feb;84(2):138-41. doi: 10.1136/adc.84.2.138. PMID 11159288
- [Background] Wiberg JM, Nordsteen J, Nilsson N. The short-term effect of spinal manipulation in the treatment of infantile colic: a randomized controlled clinical trial with a blinded observer. J Manipulative Physiol Ther. 1999 Oct;22(8):517-22. doi: 10.1016/s0161-4754(99)70003-5. PMID 10543581
- [Background] Posadzki P, Lee MS, Ernst E. Osteopathic manipulative treatment for pediatric conditions: a systematic review. Pediatrics. 2013 Jul;132(1):140-52. doi: 10.1542/peds.2012-3959. Epub 2013 Jun 17. PMID 23776117
- [Background] Dobson D, Lucassen PL, Miller JJ, Vlieger AM, Prescott P, Lewith G. Manipulative therapies for infantile colic. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004796. doi: 10.1002/14651858.CD004796.pub2. PMID 23235617